CLINICAL TRIAL: NCT01900002
Title: A Phase II Study of Sorafenib and Yttrium-90 Glass Microspheres for Advanced Hepatocellular Carcinoma, BCLC Stage C
Brief Title: Sorafenib Tosylate and Yttrium Y 90 Glass Microspheres in Treating Patients With Liver Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0870; NCI-2013-01667 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Y-90; 2012-0870 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Results first posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Advanced Adult Hepatocellular Carcinoma; BCLC Stage C Hepatocellular Carcinoma; Recurrent Adult Hepatocellular Carcinoma; Stage III Hepatocellular Carcinoma AJCC v7; Stage IIIA Hepatocellular Carcinoma AJCC v7; Stage IIIB Hepatocellular Carcinoma AJCC v7; Stage IIIC Hepatocellular Carcinoma AJCC v7; Stage IV Hepatocellular Carcinoma AJCC v7; Stage IVA Hepatocellular Carcinoma AJCC v7; Stage IVB Hepatocellular Carcinoma AJCC v7; Unresectable Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate, TheraSphere) (Experimental): Patients receive sorafenib tosylate PO BID. After 4 weeks, patients receive yttrium Y 90 glass microspheres IA. Courses of sorafenib tosylate repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Sorafenib; Drug: Sorafenib Tosylate; Radiation: Yttrium Y 90 Glass Microspheres

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Sorafenib — Given PO
  Other Names: BAY 43-9006
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib
Radiation: Yttrium Y 90 Glass Microspheres — Given IA
  Other Names: TheraSphere

SUMMARY:
This phase II trial studies how well sorafenib tosylate and yttrium Y 90 glass microspheres work in treating patients with liver cancer that cannot be removed by surgery. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Yttrium Y 90 glass microspheres use glass beads to carry radiation directly to tumor cells without harming normal cells. Giving sorafenib tosylate with yttrium Y 90 glass microspheres may be an effective treatment for liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Median progression-free survival (PFS).

SECONDARY OBJECTIVES:

I. Overall survival (OS). II. Time to radiographic progression (TTRP). III. To evaluate the safety of the combination of sorafenib (sorafenib tosylate) and Yttrium-90; adverse events (National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 [NCI-CTAE v 4.0]).

OTHER OBJECTIVES:

I. Predictive biomarkers of response to therapy and survival: will assess pre-treatment plasma level of insulin-like growth factor 1 (IGF-1) as above, and assess its predictive ability of time to progression (TTP) and OS.

OUTLINE:

Patients receive sorafenib tosylate orally (PO) twice daily (BID). After 4 weeks, patients receive yttrium Y 90 glass microspheres intra-arterially (IA). Courses of sorafenib tosylate repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to understand and be willing to sign the written informed consent form; a signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure
* Life expectancy of at least 12 weeks (3 months)
* Patients with histological or cytologically documented hepatocellular carcinoma (HCC) (documentation of original biopsy for diagnosis is acceptable if tumor tissue is unavailable) or clinical diagnosis by American Association for the Study of Liver Diseases (AASLD) criteria in cirrhotic subjects is required; for subjects without cirrhosis histological confirmation is mandatory
* Patients must have at least one tumor lesion that meets the following criteria: the lesion can be accurately measured in at least one dimension according to Response Evaluation Criteria in Solid Tumor (RECIST)
* The target lesion(s) has not been previously treated with local therapy (such as surgery, radiation therapy, hepatic arterial therapy, chemoembolization, radiofrequency ablation, percutaneous ethanol injection or cryoablation)
* Patients who have received local therapy, such as surgery, radiation therapy, hepatic arterial embolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection or cryoablation are eligible if the previously treated lesions have progressed or recurred can be identified as target lesions; local therapy must have been completed at least 4 weeks prior to the baseline scan
* Patients who have received yttrium-90 microspheres are not eligible
* Patients who have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 1
* Patients who are categorized under Barcelona-Clınic Liver Cancer (BCLC)-C stage
* Cirrhosis grade of Child-Pugh class A; Child-Pugh status should be calculated based on clinical findings and laboratory results during the screening period
* Platelet count >= 60 x 10^9/L
* Hemoglobin >= 8.5 g/dL
* Total bilirubin =< 2.5 mg/dl
* Alanine transaminase (ALT) and aspartate aminotransferase (AST) =< 5 x upper limit of normal
* Serum creatinine =< 1.5 x the upper limit of normal
* Prothrombin time (PT)-international normalized ratio (INR) =< 2.3 or PT =< 6 seconds above control
* All acute toxic effects of any prior treatment have resolved to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.0 grade 1 or less at the time of signing the informed consent form (ICF)
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug; post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 30 days after the last dose of study drug; the definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate
* Subject must be able to swallow and retain oral medication

Exclusion Criteria:

* Main portal vein thrombosis (PVT)
* Patients who are eligible for curative treatment (ablation or resection or transplantation)
* Previous or concurrent cancer other than HCC unless without evidence of disease for 5 or more years prior to entry, except cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor
* Tumor replacement > 70% of total liver volume based on visual estimation by the investigator OR tumor replacement > 50% of total liver volume in the presence of albumin < 3 mg/dL
* Contraindications to angiography and selective visceral arterial catheterization
* Any known contraindications to sorafenib including allergic reaction, pill-swallowing difficulty, uncontrolled hypertension or history of cardiac disease, significant gastrointestinal (GI) bleed within 30 days, metastatic brain disease, renal failure requiring dialysis
* Concomitant treatment or within 28 days of one of the following:

  * Any other systemic anticancer agent other than agents used for cancer prevention
  * Subjects who have used strong cytochrome P450 3A4 (CYP3A4) inducers (e.g., phenytoin, carbamazepine, phenobarbital, St. John's Wort [hypericum perforatum], dexamethasone at a dose of greater than 16 mg daily, or rifampin [rifampicin], and/or rifabutin) within 28 days before treatment
  * UDP glycosyltransferase 1 family, polypeptide A1 (UGT 1A1) and UDP glycosyltransferase 1 family, polypeptide A9 (UGT 1A9) substrates (e.g., irinotecan)
  * P-glycoprotein (Gp) substrates (e.g., Digoxin)
* Prior radiation therapy to the liver
* Prior systemic therapy for the treatment of HCC, including sorafenib
* Any history of symptomatic pulmonary compromise, such as chronic obstructive pulmonary disease
* Any prior intervention for, or ongoing compromise of, the ampulla of Vater or biliary-enteric anastomosis
* Clinically evident ascites (trace ascites on imaging is acceptable)
* Pregnant or breast-feeding patients
* A positive serum pregnancy test within 14 days prior to treatment in women of childbearing potential
* Uncontrolled hypertension (systolic pressure > 140 mm Hg or diastolic pressure > 90 mm Hg [NCI-CTCAE v4.0] on repeated measurement) despite optimal medical management
* Active or clinically significant cardiac disease including:

  * Congestive heart failure-New York Heart Association (NYHA) > class II
  * Active coronary artery disease
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin
  * Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before treatment, or myocardial infarction within 6 months before treatment
* Evidence or history of bleeding diathesis or uncontrolled coagulopathy
* Subject with any pulmonary hemorrhage/bleeding event of NCI-CTCAE v4.0 grade 2 or higher within 4 weeks before treatment; any other hemorrhage/bleeding event of NCI-CTCAE v4.0 grade 3 or higher within 4 weeks before treatment
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) within 6 months of informed consent
* Presence of a non-healing wound, non-healing ulcer, or bone fracture
* History of organ allograft. (Including corneal transplant)
* Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial
* Any malabsorption condition
* Inability to comply with the protocol and/or not willing or not available for follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09-13 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed O Kaseb, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kaseb AO, Kappadath SC, Lee SS, Raghav KP, Mohamed YI, Xiao L, Morris JS, Ohaji C, Avritscher R, Odisio BC, Kuban J, Abdelsalam ME, Chasen B, Elsayes KM, Elbanan M, Wolff RA, Yao JC, Mahvash A. A Prospective Phase II Study of Safety and Efficacy of Sorafenib Followed by 90Y Glass Microspheres for Patients with Advanced or Metastatic Hepatocellular Carcinoma. J Hepatocell Carcinoma. 2021 Sep 9;8:1129-1145. doi: 10.2147/JHC.S318865. eCollection 2021. PMID 34527608
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 2013 - December 2020. All participants were enrolled in MD Anderson
Period: Overall Study
Arm/Group | Treatment (Sorafenib Tosylate, TheraSphere)
Started | 40
Completed | 34
Not Completed | 6
Not completed — Withdrawal by Subject | 2
Not completed — ineligible for Y-90 | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Sorafenib Tosylate, TheraSphere)
Number analyzed (Participants) | 34
Age, Continuous [Mean (Full Range); unit: years] | 68.2 [48 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS)
Description: Will be monitored using the method of Thall et al. Kaplan-Meier method will be used to estimate median progression free survival (PFS) and the 95% confidence interval. Log rank test, univariate and multivariate Cox proportional hazards regression models will be used to identify prognostic factors for progression free survival (PFS).
Time Frame: From the start of therapy until failure to disease progression or death, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Sorafenib Tosylate, TheraSphere)
Number analyzed (Participants) | 34
months | 10.32 [5.78 to 14.36]

2. Secondary Outcome: Median Time to Progression (TTP)
Description: 95% credible interval will be estimated. This will be analyzed using Kaplan-Meier method, Log rank test and Cox proportional hazards regression modeling.
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Sorafenib Tosylate, TheraSphere)
Number analyzed (Participants) | 34
months | 10.38 [5.78 to 18.76]

3. Secondary Outcome: Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0
Description: To evaluate the safety of the combination of sorafenib (sorafenib tosylate) and Yttrium-90; adverse events (National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 [NCI-CTAE v 4.0]) .
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sorafenib Tosylate, TheraSphere)
Number analyzed (Participants) | 34
Participants
  Fatigue | 3
  Diarrhea | 2
  Nausea | 1
  Vomiting | 2
  Hypertension | 4
  Thrombocytopenia | 1
  Hyperbilirubinemia | 1
  Proteinuria | 1
  ALT increase | 1
  AST increase | 1

ADVERSE EVENTS:
Time Frame: adverse events were collected up to 4 years
Arm/Group | Treatment (Sorafenib Tosylate, TheraSphere)
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 11/34
Other Adverse Events (participants affected / at risk) | 27/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sorafenib Tosylate, TheraSphere) (N=34)
Dizziness (Nervous system disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Hyponatremia (Investigations) | 3
Hepatic Hemorrhage (Gastrointestinal disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Hypertenstion (Vascular disorders) | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Acute Renal Failure (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 1
Hypophosphatemia (Investigations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Rectal Bleed (Gastrointestinal disorders) | 1
Weakness (General disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sorafenib Tosylate, TheraSphere) (N=34)
Fatigue (General disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Weight Loss (Investigations) | 1
Vomiting (Gastrointestinal disorders) | 2
Palmar-Planta Erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 4
Thrombocytopenia (Investigations) | 1
Hyperbilirubinemia (Investigations) | 1
Proteinuria (Investigations) | 1
Hyponatremia (Investigations) | 1
Hypophosphatemia (Investigations) | 1
Mucositis (Gastrointestinal disorders) | 1
Encephalopathy (Nervous system disorders) | 1
ALT increase (Investigations) | 2
AST increase (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT01900002/Prot_SAP_000.pdf